CLINICAL TRIAL: NCT03849079
Title: Clinical Validation of the Inactivation Procedure for Peanut Major Allergens in the HYPONUT Product
Brief Title: Validation of the HYPONUT Product
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All prick tests are positive
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UF 7542
Record Dates: First submitted 2019-02-19; First posted 2019-02-21 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Peanut Allergy
Keywords: Peanut Allergy; Skin Prick Test; Oral Food Challenge; Hyponut
MeSH Terms: conditions — Peanut Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyponut (Experimental)
  Interventions: Other: Hyponut

INTERVENTIONS:
Other: Hyponut — Prick tests with hyponut

SUMMARY:
The HYPONUT product was previously validated in a laboratory setting ("Procédé de préparation d'aliment hypoallergénique", n° FR1250977) on 2012. A international patent was then obtained on 2013. Through the present study, the investigators would like to prove that the hypoallergenicity of the product is sustained in a clinical setting. Patients allergic to peanuts currently undergo in vivo tests to confirm their allergy: skin prick tests, and oral food challenges. In vitro tests are also performed (i.e. IgE levels for peanut and peanut components). The follow-up of patients consists in regular yearly or semestral evaluations. During one of these evaluation, the investigators will skin tests patients with the hyponut product to verify if they are sensitized to this last one as well. When skin tests will be negative, the investigators will propose to patients to take some of the product to verify its tolerability as well.

ELIGIBILITY:
Inclusion criteria:

* Patients aged more than 6
* Patients suffering from peanut allergy and followed in the Allergy Unit of the University Hospital of Montpellier (France)

Exclusion criteria:

* Pregnancy, or patients breast-feeding
* Patients treated with drugs possibly altering the results of the tests (e.g. anti-histamines)
* Patients presenting with dermographism
* Patients not fluent in French

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Skin Prick Tests evaluation | day patient enrolled

SECONDARY OUTCOMES:
Oral food challenge evaluation | day patient enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: No